CLINICAL TRIAL: NCT05498805
Title: A Randomized Controlled Phase II Trial of PD-1 Inhibitors With or Without Radiation in Patients With Advanced Melanoma
Brief Title: PD-1 Inhibitors With or Without Radiation in Advanced Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhiguo Luo, MD, PhD, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fudan-MM002
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: the Efficacy and Safety of PD-1 Inhibitors With or Without Radiotherapy in Patients With Advanced Melanoma
MeSH Terms: interventions — Radiation

STUDY DESIGN:
Intervention Model Description: radiation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): PD-1 inhibitor combined with radiotherapy, whether PD-1 inhibitor was used alone or in combination with other drugs was determined by the investigator. According to the lesion sties, SBRT or hyperfractionated radiotherapy was used.
  Interventions: Radiation: Radiation
- controlled group (Active Comparator): PD-1 inhibitor without radiotherapy, whether PD-1 inhibitor was used alone or in combination with other drugs was determined by the investigator.
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — According to the lesion sites, SBRT or hyperfractionated radiotherapy was used.

SUMMARY:
This trial was a single-center, prospective, randomized controlled phase II trial. The objective was to evaluate the efficacy and safety of PD-1 inhibitors with or without radiotherapy in patients with advanced melanoma. At the same time, tissue and peripheral blood samples of patients were collected for the determination of PD-L1 expression, ctDNA and other biomarkers and results analysis to find prognostic or curative effect predictors. A total of 92 patients were planned to be enrolled in this study.

Patients with advanced melanoma who met the inclusion criteria but did not meet the exclusion criteria were enrolled in the study and received PD-1 inhibitors with or without radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

Aged ≥18 years old, both sexes;

Malignant melanoma was confirmed by histology and pathology.

Braf, Nras, Ckit gene mutation status is unlimited.

Unresectable or metastatic melanoma, no matter lines of treatment;

Eastern Oncology Collaborative Group (ECOG) body condition score (PS) 0-2;

Predicted survival time exceeds 3 months.

Within 7 days (including 7 days) before screening, laboratory test data were used to obtain neutrophil count ≥1.5×109/L, platelet count ≥90×109/L, hemoglobin ≥90g/L (no blood transfusion within 14 days), and serum total bilirubin ≤1.25 times upper limit of normal (ULN). ALT and AST≤ 2.5 x ULN (≤ 5X ULN in patients with liver metastases); Serum creatinine ≤1.25 x ULN;

At least one radiotherapable lesion;

Subjects (or their legal representative/guardian) must sign an informed consent form stating that they understand the purpose of the study, understand the required procedures, and are willing to participate in the study.

Exclusion Criteria:

Received any investigational or antitumor drugs within 4 weeks prior to enrollment;

A history of other tumors within the past five years, except cured cervical cancer or basal cell carcinoma of the skin;

A tumor emergency that requires immediate radiotherapy, such as symptomatic brain or meningeal metastases, bone-related events, etc.

clinically significant active bleeding;

a woman who is pregnant or breastfeeding; Persons who are fertile but do not take adequate contraceptive measures;

Alcoholism or drug addiction;

with active, or have a history and are likely to relapse of patients with autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerular inflammation, etc.), or high risk (e.g., received organ transplants on immunosuppressive therapy) of the patients. Exceptions are autoimmune hypothyroidism that requires only hormone replacement therapy or skin conditions that do not require systemic treatment.

patients who required systemic treatment with corticosteroids (doses equivalent to > 10mg prednisone/day) or other immunosuppressive agents within 14 days prior to enrollment or during the study. Use topical or inhaled glucocorticoids, or short-term (≤7 days) glucocorticoids for the prevention or treatment of non-autoimmune, infrequently occurring allergic diseases.

Critical organ failure or other serious disease, including interstitial pneumonia, clinically relevant coronary disease, cardiovascular disease, or a history of myocardial infarction, congestive heart failure, unstable angina, symptomatic pericardial effusion, or unstable arrhythmia in the 6 months prior to enrollment;

Have a history of human immunodeficiency virus infection, another acquired or congenital immunodeficiency disease, or a history of organ transplantation, or stem cell transplantation;

A patient with active chronic hepatitis B or active hepatitis C. HBV carriers, medically stable hepatitis B (DNA titer ≤103 copies /ml), and cured hepatitis C (HCV RNA negative) patients were eligible for enrollment.

A history of severe neurological or psychiatric problems; Severe infection; Active disseminated intravascular coagulation or other comorbidities that, in the investigator's judgment, seriously compromise patient safety or interfere with study completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2022-08-15 (Estimated); Primary Completion 2024-10-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 7 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cencer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided